CLINICAL TRIAL: NCT05427500
Title: Stellate Ganglion Block in the Treatment of Posttraumatic Stress Disorder: Outcome Evaluation, Mechanism of Action, and Integration in Care - A Phase III Randomized Controlled Trial
Brief Title: Stellate Ganglion Block in the Treatment of Posttraumatic Stress Disorder
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: The Royal's Institute of Mental Health Research (Other)
Collaborators: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Rebecca Gomez, MD, Psychiatrist, The Royal's Institute of Mental Health Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022001
Record Dates: First submitted 2022-06-09; First posted 2022-06-22 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: PTSD
Keywords: Stellate Gangllion Block; Canadian Armed Forces; Veterans; Royal Canadian Mounted Police
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single SGB (Other): This arm will receive a single 5 mL dose of 0.5% preservative-free bupivacaine.
  Interventions: Drug: 5 mL of 0.5% preservative-free bupivacaine
- Repeated SGB (Other): This arm will receive two 5 mL doses of 0.5% preservative-free bupivacaine.
  Interventions: Drug: 5 mL of 0.5% preservative-free bupivacaine

INTERVENTIONS:
Drug: 5 mL of 0.5% preservative-free bupivacaine — IV will be inserted. Patient will be connected to cardiorespiratory monitors. The neck will be cleansed twice. A high frequency (15-6 MHz) linear ultrasound probe will be used to identify the arteries, jugular vein, and other important vasculature. Once a clear path for the needle is identified, the skin is anesthetized. A cutting tip spinal needle is then inserted at the lateral aspect of the field and advanced in-plane under ultrasound visualization. A test injection is injected to verify placement, then 5 mL of 0.5% preservative-free bupivacaine will be injected. Per standard SGB procedure, vitals will be measured post-SGB and participants will remain in the clinic for approximately 15 minutes to monitor for any serious adverse events.
  Other Names: SteriMax Bupivicaine

SUMMARY:
The most common treatment for Posttraumatic Stress Disorder (PTSD) is trauma-focused therapy and/or prescription of medication(s). However, these treatments may not directly reduce symptoms associated with PTSD, making it difficult for patients to be treated for this condition and recover. Stellate ganglion block (SGB) is a medical procedure that involves injection of a local anesthetic (a medication that causes reduced sensation/feeling in a given area) around the stellate ganglion, which is a collection of nerves near the base of the neck. This procedure causes a short-lived, temporary shutdown of nerve signals (up to 5-7 hours) and is commonly performed in Canada for certain pain and medical conditions. In the last decade, several studies, including those involving members of military groups, have shown that SGB can result in a rapid and sustained drop in symptoms related to PTSD such as overwhelming anxiety, increased irritability, heightened alertness, and exaggerated startle. Considering these results and the known safety of this procedure (as demonstrated by previous research and use in other illnesses), SGB has been increasingly used to treat PTSD among veterans in the United States but has not yet been evaluated in Canada. More research is thereby needed to use SBG as a method of PTSD treatment in Canada, and to better understand how it works to reduce symptoms associated with this condition. Health Canada, the organization which oversees clinical trials such as this one, has not approved the use of the SGB procedure for PTSD in the general population, however Health Canada has allowed the use of SGB in this study to better understand how it works and how it may be used in the future to treat PTSD-related symptoms in those who feel that common treatments are not effective.

DETAILED DESCRIPTION:
Posttraumatic Stress Disorder (PTSD) is a trauma- and stress-related disorder arising from an experienced or witnessed traumatic event, most commonly actual or threatened death, serious injury, or sexual violence. There is a distinct pattern of intrusion and avoidance, as well as negative alterations in cognitions, mood, arousal, and reactivity, leading to serious impairments in personal, social and occupational functioning. The risk of PTSD is elevated in military and public safety personnel, and first responders. Despite advances in evidence-based treatments for PTSD, optimal outcomes are often not achieved, particularly in military veterans. One of the treatment-interfering factors is persistent hyperarousal (abnormally heightened state of anxiety and alertness), which prevents engagement in trauma processing and contributes to medication intolerance and substance misuse. The search for novel methods to target hyperarousal and underlying responses of the sympathetic nervous system have provided some promising pharmacologic approaches, such as the use of the adrenergic (adrenaline-related) blockers propranolol and prazosin. There is a need for novel and complementary approaches to normalize sympathetic (fight-or-flight) regulation in PTSD to provide symptom relief and facilitate its treatment and recovery.

Stellate ganglion block (SGB) is a medical procedure that involves injection of local anesthetic around the stellate ganglion, which is a collection of sympathetic (fight-or-flight) nerves near the base of the neck (C6-7). This procedure causes a short-lived shutdown of sympathetic nerve signals (up to 5-7 hours) and is commonly performed in Canada for certain pain and medical conditions. SGB is an interventional procedure that temporarily blocks sympathetic signaling to the arms, neck and head with long-established therapeutic benefits for sympathetically maintained pain and other medical conditions. In the past decade, SGB was found to provide a rapid and sustained reduction of PTSD symptoms in numerous case reports and series. Further, two randomized controlled trials of SGB in PTSD have been conducted. The first study in active and retired military personnel with combat and non-combat PTSD did not differentiate the effect of SGB from sham control one week or one month post-injection , although these results were inconclusive due to methodological limitations. The second study in active-duty military personnel established substantial efficacy of SGB that was administered twice in a 2-week interval when assessed at eight weeks after the first injection . Notably, most of the studies above were conducted in predominantly male active-duty military samples and none specifically in veterans, law enforcement officers, or first responders. Considering these results and the known safety of this procedure, SGB has been increasingly used to treat PTSD in the United States Veterans Affairs (VA) system, but has not yet been evaluated in Canada.

The mechanism of action of SGB in PTSD is not well understood. Presumably, SGB directly reduces peripheral sympathetic tone but may also project to the central nervous system to activate neuroplasticity processes. The current consensus is that SGB has a unique adjunct potential in PTSD treatment, but the parameters of its use and mechanism of action require further study. In order to enhance care and in response to requests from our patients and their clinicians, we initiated a collaboration between the OSI and TOH Pain clinics to facilitate access to SGB for our patients, particularly those who are not improving with traditional therapies because of intractable hyperarousal and anxiety. To date, 15 patients have undergone off-label SGB procedures at The Ottawa Hospital (TOH) Pain Clinic, seven for whom we have clinical data up to eight weeks post-SGB. We are still collecting follow-up data for the other eight patients, who had the procedure done more recently. Of those seven who underwent SGB procedures prior to October 2021, five were responders on the PTSD Checklist for DSM-5 (PCL-5), as evidenced by a 10-point decrease in the total score, between one week pre-SGB and eight weeks post-SGB. Mean Quick Inventory of Depressive Symptomatology (QIDS-SR) scores decreased from the severe to moderate range. Within 2 weeks of the procedure, one patient commented that he had "less anxiety, no panic attacks," and another reported, "It was like the entire planet felt less menacing and I felt calmer than I had in years." There were no serious adverse events related to the SGB procedure. In summary, current treatments for PTSD have shortcomings and less success in military veterans. One of the most significant challenges for recovery from PTSD is an overactive "fight-or-flight" state, fueled by the sympathetic nervous system. Patients struggle with near constant hyperarousal as they are in a state of physical and mental readiness to react to a threat. While this reaction is appropriate in dangerous situations, as a symptom of PTSD, it becomes excessive and uncontrollable, leading to persistent anxiety, irritability, agitation, startle, and sleep problems as well as triggering traumatic memories and standing in the way of regular life activities. Currently, even the best treatments for PTSD do not directly reduce hyperarousal or sympathetic activity, making it more difficult for patients to engage in and benefit from trauma-focused therapy or medications. Sufferers are often prompted to self-medicate with alcohol and other substances, which also negatively impact the patient's family and support network. This significant treatment gap calls for exploring novel ways to lessen the entrenched "fight or flight" state in those with PTSD.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of PTSD according to DSM-5 criteria with prominent and persistent cluster E hyperarousal symptoms
2. Age 18-69 years
3. Under care of a mental health clinician
4. Not benefited from adequate trials of pharmacological or psychological evidence-based treatment and/or a preference and consent for a trial of SGB

Exclusion Criteria:

1. Assessed with high risk for suicide in the last 30 days (per patient's treating clinician at OSI clinic)
2. Diagnosis of bipolar or psychotic disorder
3. Moderate to severe substance use within the last 30 days (based on chart and verbal report from patient)
4. In process of disability assessment or legal action
5. Moderate or severe TBI (based on chart and verbal report from patient)
6. Pregnancy or breastfeeding
7. Current anticoagulant use (eligible if can be held before the procedure)
8. History of bleeding disorder (based on chart and verbal report from patient)
9. Infection, mass or anatomic abnormalities at target injection site
10. Myocardial infarction within 6 months of procedure (based on chart and verbal report from patient)
11. Pathologic bradycardia or irregularities of heart rate or rhythm (based on chart and verbal report from patient)
12. Symptomatic hypotension (BP<90/60 + clinical symptoms of hypotension)
13. Phrenic or laryngeal nerve palsy (based on chart and verbal report from patient)
14. History of glaucoma (based on chart and verbal report from patient)
15. Uncontrolled seizure disorder (based on chart and verbal report from patient)
16. Known history of allergy to local anesthetics (based on chart and verbal report from patient)
17. Severe COPD (based on chart and verbal report from patient)
18. Pneumothorax (based on chart and verbal report from patient)
19. Contralateral pneumonectomy or non-functional lung (based on chart and verbal report from patient)
20. Active systemic infection (based on chart and verbal report from patient)
21. Patient refusal/inability to tolerate procedure/positioning
22. Contraindication to MR imaging
23. Any other condition that in the opinion of the investigator could create a hazard to the participant's safety, endanger the study procedures, or interfere with the interpretation of study results.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-03-30 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Monitoring patient response and remission of PTSD symptoms | From pre-SGB to final study visit 12-weeks post procedure.
  Proportion of patients showing response (at least 10-point reduction) and remission (total score < 33) in symptoms of PTSD on PCL-5
Monitoring patient improvement on Clinician Administered PTDS Scale for DSM-5 (CAPS-5) | From pre-SGB to final study visit 12-weeks post procedure.
  Proportion of patients showing response (at least 10-points reduction) and loss of diagnosis on CAPS-5
Monitoring patient improvement in symptom burden and functioning | From pre-SGB to final study visit 12-weeks post procedure.
  Proportion of patients achieving reliable change (at least 14-point reduction) in the total score on OQ45.2 reflecting improvement in symptom burden and functioning

SECONDARY OUTCOMES:
Changes from baseline in hypervigilance | From pre-SGB to final study visit 12-weeks post procedure.
  Measured by the Brief Hypervigilance Scale
Changes from baseline in anxiety | From pre-SGB to final study visit 12-weeks post procedure.
  Measured by the Overall Anxiety Severity Impairment Scale
Changes from baseline in depression | From pre-SGB to final study visit 12-weeks post procedure.
  Measured by the Quick Inventory of Depressive Symptomatology
Changes from baseline in pain scale scores | From pre-SGB to final study visit 12-weeks post procedure.
  Measured by the Brief Pain Inventory
Ratings of participant satisfaction and recommendations for future use of SGB | From pre-SGB to final study visit 12-weeks post procedure.
  Measured by qualitative self report scale
Changes in participant's symptomatology and overall functioning from the perspective of the participant's family and support network | From pre-SGB to final study visit 12-weeks post procedure.
  Measured by Family And Support Team-Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gomez, MD, Principal Investigator — Psychiatrist at the OSI Clinic at the Royal Ottawa Mental Health Centre
Locations (1):
- The Royal Ottawa Mental Health Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Psychiatric Association, DSM-5 Task Force. (2013). Diagnostic and Statistical Manual of Mental Disorders: DSM-5™ (5th ed.). American Psychiatric Publishing, Inc
- [Background] Steenkamp MM, Litz BT, Hoge CW, Marmar CR. Psychotherapy for Military-Related PTSD: A Review of Randomized Clinical Trials. JAMA. 2015 Aug 4;314(5):489-500. doi: 10.1001/jama.2015.8370. PMID 26241600
- [Background] Krystal JH, Davis LL, Neylan TC, A Raskind M, Schnurr PP, Stein MB, Vessicchio J, Shiner B, Gleason TC, Huang GD. It Is Time to Address the Crisis in the Pharmacotherapy of Posttraumatic Stress Disorder: A Consensus Statement of the PTSD Psychopharmacology Working Group. Biol Psychiatry. 2017 Oct 1;82(7):e51-e59. doi: 10.1016/j.biopsych.2017.03.007. Epub 2017 Mar 14. No abstract available. PMID 28454621
- [Background] Hoge CW. Interventions for war-related posttraumatic stress disorder: meeting veterans where they are. JAMA. 2011 Aug 3;306(5):549-51. doi: 10.1001/jama.2011.1096. No abstract available. PMID 21813436
- [Background] DePierro J, Lepow L, Feder A, Yehuda R. Translating Molecular and Neuroendocrine Findings in Posttraumatic Stress Disorder and Resilience to Novel Therapies. Biol Psychiatry. 2019 Sep 15;86(6):454-463. doi: 10.1016/j.biopsych.2019.07.009. Epub 2019 Jul 24. PMID 31466562
- [Background] Aleanakian R, Chung BY, Feldmann RE Jr, Benrath J. Effectiveness, Safety, and Predictive Potential in Ultrasound-Guided Stellate Ganglion Blockades for the Treatment of Sympathetically Maintained Pain. Pain Pract. 2020 Jul;20(6):626-638. doi: 10.1111/papr.12892. Epub 2020 May 17. PMID 32255250
- [Background] Lipov EG, Joshi JR, Lipov S, Sanders SE, Siroko MK. Cervical sympathetic blockade in a patient with post-traumatic stress disorder: a case report. Ann Clin Psychiatry. 2008 Oct-Dec;20(4):227-8. doi: 10.1080/10401230802435518. No abstract available. PMID 19034755
- [Background] Mulvaney SW, Lynch JH, Hickey MJ, Rahman-Rawlins T, Schroeder M, Kane S, Lipov E. Stellate ganglion block used to treat symptoms associated with combat-related post-traumatic stress disorder: a case series of 166 patients. Mil Med. 2014 Oct;179(10):1133-40. doi: 10.7205/MILMED-D-14-00151. PMID 25269132
- [Background] Lipov E, Ritchie EC. A review of the use of stellate ganglion block in the treatment of PTSD. Curr Psychiatry Rep. 2015 Aug;17(8):599. doi: 10.1007/s11920-015-0599-4. PMID 26073361
- [Background] Hanling SR, Hickey A, Lesnik I, Hackworth RJ, Stedje-Larsen E, Drastal CA, McLay RN. Stellate Ganglion Block for the Treatment of Posttraumatic Stress Disorder: A Randomized, Double-Blind, Controlled Trial. Reg Anesth Pain Med. 2016 Jul-Aug;41(4):494-500. doi: 10.1097/AAP.0000000000000402. PMID 27187898
- [Background] Rae Olmsted KL, Bartoszek M, Mulvaney S, McLean B, Turabi A, Young R, Kim E, Vandermaas-Peeler R, Morgan JK, Constantinescu O, Kane S, Nguyen C, Hirsch S, Munoz B, Wallace D, Croxford J, Lynch JH, White R, Walters BB. Effect of Stellate Ganglion Block Treatment on Posttraumatic Stress Disorder Symptoms: A Randomized Clinical Trial. JAMA Psychiatry. 2020 Feb 1;77(2):130-138. doi: 10.1001/jamapsychiatry.2019.3474. PMID 31693083
- [Background] Peterson K, Bourne D, Anderson J, Mackey K, Helfand M. Evidence Brief: Effectiveness of Stellate Ganglion Block for Treatment of Posttraumatic Stress Disorder (PTSD) [Internet]. Washington (DC): Department of Veterans Affairs (US); 2017 Feb. Available from http://www.ncbi.nlm.nih.gov/books/NBK442253/ PMID 28742302